CLINICAL TRIAL: NCT03584217
Title: Renal HEIR Study: Renal Hemodynamics, Energetics and Insulin Resistance in Youth Onset Type 2 Diabetes Study
Acronym: Renal-HEIR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-1752
Record Dates: First submitted 2018-06-28; First posted 2018-07-12 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Nephropathy; Adolescent Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Kidney Diseases; Pediatric Obesity | interventions — p-Aminohippuric Acid; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clinical Investigation (Other): All participants will undergo GFR (Iohexol Inj 300 MG/ML), ERPF (Aminohippurate Sodium Inj 20%) in addition to renal BOLD and ASL MRI.
  Interventions: Drug: Aminohippurate Sodium Inj 20%; Drug: Iohexol Inj 300 MG/ML; Procedure: Renal Biopsy

INTERVENTIONS:
Drug: Aminohippurate Sodium Inj 20% — Diagnostic aid/agent used to measure effective renal plasma flow (ERPF)
  Other Names: Sodium 4-amino hippurate (PAH) inj 20% 2g/10mL; Para-aminohippurate; Aminohippuric acid
Drug: Iohexol Inj 300 MG/ML — Diagnostic aid/agent used to measure glomerular filtration rate (GFR)
  Other Names: omnipaque 300
Procedure: Renal Biopsy — Minimally invasive outpatient procedure in interventional radiology to obtain renal tissue cores.
  Other Names: Kidney Biopsy

SUMMARY:
Type 2 diabetes (T2D) in youth is increasing in prevalence in parallel with the obesity epidemic. In the US, almost half of patients with renal failure have DKD, and ≥80% have T2D. Compared to adult-onset T2D, youth with T2D have a more aggressive phenotype with greater insulin resistance (IR), more rapid β-cell decline and higher prevalence of diabetic kidney disease (DKD), arguing for separate and dedicated studies in youth-onset T2D. Hyperfiltration is common in youth with T2D, and predicts progressive DKD. Hyperfiltration may also be associated with early changes in intrarenal hemodynamic function, including increased renal plasma flow (RPF) and glomerular pressure. Despite the high prevalence and gravity of DKD in youth-onset T2D, widely effective therapeutic options are lacking. The investigators' preliminary data support a strong association between IR and hyperfiltration in youth-onset T2D, but the pathology contributing to this relationship remains unclear. A better understanding of the pathophysiology underlying hyperfiltration and its relationship with IR is critical to inform development of new therapeutics. The investigators' overarching hypotheses are that: 1) hyperfiltration in youth-onset T2D is associated with changes in intrarenal hemodynamics, resulting in increased renal oxygen demand, 2) the demand is unmet by the inefficient fuel profile associated with IR (decreased glucose oxidation and increase free fatty acid [FFA] oxidation), resulting in renal hypoxia and ultimately renal damage. To address these hypotheses, the investigators will measure peripheral insulin sensitivity, adipose insulin sensitivity (FFA suppression), glomerular filtration rate (GFR), RPF, and renal oxygenation in youth with T2D (n=60), obesity (n=20) and in lean (n=20) controls. To further investigate the mechanisms of renal damage in youth with T2D, two optional procedures are included in the study: 1) kidney biopsy procedure and 2) induction of induced pluripotent stem cells (iPSCs) to assess morphometrics and genetic expression of renal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Obese youth with and without T2D (≥54 kg) and lean controls
* Age 12-21 years
* Weight <300 lbs., no implanted metal devices
* HbA1c < 11% and no recent diabetic ketoacidosis or hyperosmolar hyperglycemia
* No anemia
* BMI >5th percentile for lean controls

Exclusion Criteria:

* T2D onset (diagnosis) > 18 years of age
* Prepubertal
* eGFR <60ml/min/1.73m2 or creatinine > 1.5mg/dl or history of ACR≥300mg/g
* ACE inhibitors, angiotensin receptor blockers (ARB), diuretics, sodium-glucose co-transport (SGLT) 2 or 1 blockers, daily NSAIDs or aspirin, sulfonamides, procaine, thiazosulfone or probenecid.
* Seafood or iodine allergy
* Pregnancy
* MRI scanning contraindications (claustrophobia, implantable devices, >300 lbs)

Additional exclusion criteria for participants undergoing optional kidney biopsy:

* Evidence of bleeding disorder or complications from bleeding
* Use of aspirin, NSAIDS or other blood thinner that cannot be safely stopped for a sufficient time period before and after the biopsy so as to add no additional risk of bleeding
* Blood urea nitrogen (BUN) > 80 gm/dL
* INR > 1.4
* PTT > 35 seconds
* Hemoglobin (Hgb) < 10 mg/dL
* Platelet count < 100,000 / µL
* Uncontrolled or difficult to control hypertension (> 150/90 mmHg at the day of biopsy)
* eGFR < 40 mL/min/1.73m2
* Single kidney (either by history, documented by prior imaging or ultrasound performed prior to the biopsy)
* > 2 cm discrepancy between left and right kidney sizes based on largest longitudinal diameter determined by ultrasound performed prior to the biopsy.
* Kidney size: One or both kidneys < 9 cm
* Hydronephrosis or other important renal ultrasound findings such as significant stone disease
* Any evidence of a current urinary tract infection as indicated on day of biopsy
* Clinical evidence of non-diabetic renal disease
* Positive urine pregnancy test or pregnancy

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Effective renal plasma flow (ERPF) | 4 hours
  Measured by PAH clearance
Glomerular filtration rate (GFR) | 4 hours
  Measured by iohexol clearance

SECONDARY OUTCOMES:
Insulin sensitivity | 4 hours
  Measured by hyperinsulinemic-euglycemic clamp
Renal oxygenation | 60 min
  Blood oxygen level dependent (BOLD) MRI
Renal perfusion | 10 min
  Arterial spin labeling (ASL) MRI

OTHER OUTCOMES:
Podocyte numerical density and number per glomerulus | 4 hours
  Measured by light microscopy from tissue obtained by renal biopsy
Foot process width of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Detachment and endothelial fenestration of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Podocyte volume of glomeruli | 4 hours
  Measured by electron microscopy from tissue obtained by renal biopsy
Number and identity of RNA in kidney cells | 4 hours
  Measured from tissue obtained by renal biopsy
Epigenetic profiling | 4 hours
  Measured from tissue obtained by renal biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Petter Bjornstad, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vigers T, Vinovskis C, Li LP, Prasad P, Heerspink H, D'Alessandro A, Reisz JA, Piani F, Cherney DZ, van Raalte DH, Nadeau KJ, Pavkov ME, Nelson RG, Pyle L, Bjornstad P. Plasma levels of carboxylic acids are markers of early kidney dysfunction in young people with type 1 diabetes. Pediatr Nephrol. 2023 Jan;38(1):193-202. doi: 10.1007/s00467-022-05531-3. Epub 2022 May 4. PMID 35507146
- [Derived] Vinovskis C, Li LP, Prasad P, Tommerdahl K, Pyle L, Nelson RG, Pavkov ME, van Raalte D, Rewers M, Pragnell M, Mahmud FH, Cherney DZ, Johnson RJ, Nadeau KJ, Bjornstad P. Relative Hypoxia and Early Diabetic Kidney Disease in Type 1 Diabetes. Diabetes. 2020 Dec;69(12):2700-2708. doi: 10.2337/db20-0457. Epub 2020 Jul 31. PMID 32737116